CLINICAL TRIAL: NCT03169660
Title: Efficacy of Intravitreal Aflibercept Monotherapy for Submacular Hemorrhage Secondary to Neovascular Age-Related Macular Degeneration: A Prospective Clinical Trial
Brief Title: Intravitreal Aflibercept for Submacular Hemorrhage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kim's Eye Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Jae Hui Kim, M.D., Kim's Eye Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-2014-032
Record Dates: First submitted 2015-09-02; First posted 2017-05-30 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Exudative Age-related Macular Degeneration
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment group (Experimental): Eyes with submacular hemorrhage secondary to exudative age-related macular degeneration and were treated with vascular endothelial growth factor trap-eye.
  Interventions: Drug: Vascular endothelial growth factor trap-eye

INTERVENTIONS:
Drug: Vascular endothelial growth factor trap-eye — Intravitreal injection of vascular endothelial growth factor trap-eye During the first 3 months, 3 monthly injections are performed After 3 serial injections, additional injections are performed once per 2 months until 48 weeks after the initial injection.
  Other Names: Eylea

SUMMARY:
The prognosis of exudative age-related macular degeneration (AMD) accompanied by submacular hemorrhage is generally poor. A recently developed anti-VEGF agent eyeliaTM is also a useful treatment option for exudative AMD. However, one major limitation of VIEW study was that lack of data regarding eyes with submacular hemorrhage. The purpose of the present study was to evaluate the efficacy of Eylea in submacular hemorrhage secondary to exudative AMD.

DETAILED DESCRIPTION:
The prognosis of exudative age-related macular degeneration (AMD) accompanied by submacular hemorrhage is generally poor. Although anti-vascular endothelial growth factor (VEGF) has been demonstrated excellent efficacy in the treatment of exudative AMD, eyes with submacular hemorrhage were excluded from the previous well-known clinical trials. The exclusion of these patients may probably be determined by some concerns suggesting possible poor prognosis in these patients. Firstly, it was well known that subretinal hemorrhage itself induces retinal damage and degeneration. Secondly, it was not certain whether the drug penetrates through hemorrhage and stabilize to the underlying lesion or not. As a result, the efficacy in submacular hemorrhage could not be demonstrated in these clinical trials.

The efficacy of anti-VEGF therapy in eyes with submacular hemorrhage has recently been spotlighted. Several reports demonstrated significant improvement in visual acuity after anti-VEGF monotherapy, including LucentisTM, AvastinTM, or both, in eyes with exudative AMD with submacular hemorrhage. Although histopathologic evidence using animal model has not been presented, results of these clinical studies suggest that anti-VEGF may penetrates the hemorrhage and stabilize the underlying lesion. Recently, a large prospective clinical trial that evaluated the efficacy of anti-VEGF therapy in this condition showed favorable outcome. Result of this study may be published in a near future

A recently developed anti-VEGF agent eyeliaTM is also a useful treatment option for exudative AMD. The result of VIEW study clearly demonstrated that this new agent has comparable efficacy to LucentisTM using less frequent injection schedule. However, one major limitation of VIEW study was that lack of data regarding eyes with submacular hemorrhage. Investigators carefully reviewed the study protocol of VIEW study and found that lesions composed of >50% blood were excluded. In addition, investigators could not aware any report in English literature that evaluated the efficacy of eyeliaTM in exudative AMD with submacular hemorrhage.

It took almost 8 years to demonstrate the efficacy of two previously available anti-VEGF agents (LucentisTM and AvastinTM) in eyes with submacular hemorrhage. Investigators believe that a prospective study evaluating the efficacy of eyeliaTM in exudative AMD with submacular hemorrhage may help to achieve a consensus that eyeliaTM is also a useful treatment for submacular hemorrhage within a relatively short time.

The purpose of the present study was to evaluate the efficacy of Eylea in submacular hemorrhage secondary to exudative AMD.

ELIGIBILITY:
Inclusion Criteria:

1. 50 years of older
2. Newly diagnosed, treatment-naïve exudative AMD
3. Fovea-involving submacular hemorrhage greater than 1 disc areas at diagnosis

Exclusion Criteria:

1. History of previous treatment for neovascular AMD
2. Greater than 15 disc diameter areas of hemorrhage extent
3. History of vitreoretinal surgery
4. History of glaucoma surgery, such as trabeculectomy or glaucoma implant surgery
5. History of ocular steroid injection therapy within 1 month
6. History of cataract surgery within 3 months
7. Aphakia or anterior chamber intraocular lens implantation
8. Spherical equivalents greater than -6.0 diopters
9. evidence of other retinal disorders that may affect visual function including diabetic retinopathy, hypertensive retinopathy, epiretinal membrane, macular hole, and microaneurysm
10. severe media opacity
11. uncontrolled systemic disorders, including hypertension or diabetes mellitus
12. history of major systemic vascular events, such as myocardial infarction and stroke
13. hypersensitivity to aflibercept
14. ocular or periocular infection
15. active intraocular inflammation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2019-01-20 (Actual)

PRIMARY OUTCOMES:
Changes in Early Treatment of Diabetic Retinopathy Study visual acuity Score | Changes from baseline in visual acuity at 56 weeks
  Increase or decrease in the Early Treatment of Diabetic Retinopathy Study letter score

SECONDARY OUTCOMES:
Proportion of patients who exhibited 15 letters or greater change in visual acuity | 56 weeks
  Changes in visual acuity of 15 Early Treatment Diabetic Retinopathy Study (ETDRS) letters or greater
Changes in central macular thickness | Changes from baseline in central macular thickness at 56 weeks
  Changes in central macular thickness (1 mm diameter centered at the centered at the fovea which is measured by optical coherence tomography)
Duration of complete hemorrahge resolution | 56 weeks
  Duration between the first injection and the complete hemorrhage resolution
Incidence of recurrence of submacular hemorrhage or fluid | 56 weeks
  New development or increase in the amount of hemorrhage or fluid
Leakage on angiography | 56 week
  Leakage on angiography

CONTACTS AND LOCATIONS:
Overall Officials: Jong Woo Kim, M.D., Principal Investigator — Kim's Eye Hospital, Seoul, South Korea
Locations (1):
- Kim's Eye Hospital, Seoul, South Korea